CLINICAL TRIAL: NCT00716625
Title: Special Investigation For RCC Of Sutent (Regulatory Post Marketing Commitment Plan).
Brief Title: Special Investigation For Renal Cell Carcinoma (RCC) Of Sunitinib Malate (Regulatory Post Marketing Commitment Plan)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6181176
Record Dates: First submitted 2008-07-15; First posted 2008-07-16 (Estimated); Results first posted 2017-01-18 (Estimated); Last update posted 2023-05-03 (Actual); Status verified 2016-11

CONDITIONS: Carcinoma, Renal Cell
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- sunitinib malate: Patients taking sunitinib malate
  Interventions: Drug: sunitinib malate

INTERVENTIONS:
Drug: sunitinib malate — SUTENT® Capsule 12.5 mg, depending on the Investigator prescription. Frequency and duration are according to Package Insert as follows. "The usual adult dosage for oral sunitinib is 50 mg once daily, 4 weeks on followed by 2 weeks off (Schedule 4/2). This comprises 1 treatment cycle, which may be repeated.
  The dosage may be decreased according to the patient's clinical condition."
  Other Names: Sutent

SUMMARY:
The objective of this surveillance is to collect information about 1) adverse drug reaction not expected from the LPD (unknown adverse drug reaction), 2) the incidence of adverse drug reactions in this surveillance, and 3)factors considered to affect the safety and/or efficacy of this drug.

DETAILED DESCRIPTION:
All the patients whom an investigator prescribes the first sunitinib malate(Sutent) should be registered.

ELIGIBILITY:
Inclusion Criteria:

* Patients need to be administered sunitinib malate (Sutent) in order to be enrolled in the surveillance.

Exclusion Criteria:

* Patients not administered sunitinib malate (Sutent).

Min Age: 0 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients whom an investigator involving A6181176 prescribes the sunitinib malate (Sutent).
Sampling Method: Probability Sample
Enrollment: 1674 (Actual)
Dates: Start 2008-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181176&StudyName=Special%20Investigation%20For%20Renal%20Cell%20Carcinoma%20%28RCC%29%20Of%20Sunitinib%20Malate%20%28Regulatory%20Post%20Marketing%20Commitment%20Plan%29

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib Malate: Usually, 50 mg of sunitinib malate was orally administered to adult participants once daily in repetitive cycles of 4 weeks on treatment followed by 2 weeks off according to Japanese package insert.
Period: Overall Study
Arm/Group | Sunitinib Malate
Started | 1674
Completed | 1673
Not Completed | 1
Not completed — Safety was not Assessable | 1

BASELINE CHARACTERISTICS:
Population: In total, 1674 participants were enrolled in the study. Of the 1674 participants, 1 participant was excluded from the baseline analysis because the safety was not assessable.
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 1673
Age, Customized [Number; unit: Participants]
  <15 years | 1
  >=15 and <65 years | 940
  ˃=65 years | 712
  Unknown | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 421
  Male | 1252

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Related Adverse Events
Description: A treatment-related adverse event was any untoward medical occurrence attributed to sunitinib malate in a participant who received sunitinib malate. Relatedness to sunitinib malate was assessed by the investigator and sponsor (Pfizer Japan Inc.).
Time Frame: MAX 2 Years
Population: Safety analysis set comprised of participants who had met the inclusion criteria and had received sunitinib malate at least once.
Measure: Number; unit: Participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 1673
Participants | 1599 [19.5 to 23.8]

2. Primary Outcome: Objective Response Rate
Description: Percentage of participants with objective response per Response Evaluation Criteria In Solid Tumors Criteria (RECIST V1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR),>=30% decrease in the sum of the longest diameter of target lesion; Overall Response(OR) = CR + PR. The result was presented along with the corresponding exact 2-sided 95% confidence interval (CI).
Time Frame: MAX 2 Years
Population: Efficacy analysis set comprised of participants in safety analysis set who had efficacy evaluation.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 1430
Percentage of participants | 21.9 [19.8 to 24.1]

3. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events in Pediatric Population
Description: A treatment-related adverse event was any untoward medical occurrence attributed to sunitinib malate in a participant who received sunitinib malate. Relatedness to sunitinib malate was assessed by the investigator and sponsor (Pfizer Japan Inc.). Pediatric population was defined as the participants who aged younger than 15, and adult population was defined as those aged 15 or older.
Time Frame: MAX 2 Years
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- Pediatric: Participants aged ˂15 years who received sunitinib malate according to Japanese package insert
- Adult: Participants aged ˃=15 years who received sunitinib malate according to Japanese package insert
- Unknown: Participants with unknown age who received sunitinib malate according to Japanese package insert
Arm/Group | Pediatric | Adult | Unknown
Number analyzed (Participants) | 1 | 1652 | 20
Participants | 1 [19.5 to 23.8] | 1581 | 17

4. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events in Elderly Population
Description: A treatment-related adverse event was any untoward medical occurrence attributed to sunitinib malate in a participant who received sunitinib malate. Relatedness to sunitinib malate was assessed by the investigator and sponsor (Pfizer Japan Inc.). Elderly population was defined as the participants who aged 65 or older.
Time Frame: MAX 2 Years
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- Elderly: Participants aged ˃=65 years who received sunitinib malate according to Japanese package insert
- Non-elderly: Participants aged ˂65 years who received sunitinib malate according to Japanese package insert
Arm/Group | Elderly | Non-elderly | Unknown
Number analyzed (Participants) | 712 | 941 | 20
Participants | 688 [19.5 to 23.8] | 894 | 17

5. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events Who Had Hepatic Impairment
Description: A treatment-related adverse event was any untoward medical occurrence attributed to sunitinib malate in a participant who received sunitinib malate. Relatedness to sunitinib malate was assessed by the investigator and sponsor (Pfizer Japan Inc.). Hepatic impairment referred not to transient laboratory test value abnormalities, but to the events that were clinically noteworthy and required follow-up.
Time Frame: MAX 2 Years
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- With Hepatic Impairment: Participants with baseline hepatic impairment who received sunitinib malate according to Japanese package insert
- Without Hepatic Impairment: Participants without baseline hepatic impairment who received sunitinib malate according to Japanese package insert
- Unknown: Participants with no information on baseline hepatic impairment who received sunitinib malate according to Japanese package insert
Arm/Group | With Hepatic Impairment | Without Hepatic Impairment | Unknown
Number analyzed (Participants) | 162 | 1506 | 5
Participants | 154 [19.5 to 23.8] | 1441 | 4

6. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events Who Had Renal Impairment
Description: A treatment-related adverse event was any untoward medical occurrence attributed to sunitinib malate in a participant who received sunitinib malate. Relatedness to sunitinib malate was assessed by the investigator and sponsor (Pfizer Japan Inc.). Renal impairment referred not to transient laboratory test value abnormalities, but to the events that were clinically noteworthy and required follow-up.
Time Frame: MAX 2 Years
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- With Renal Impairment: Participants with baseline renal impairment who received sunitinib malate according to Japanese package insert
- Without Renal Impairment: Participants without baseline renal impairment who received sunitinib malate according to Japanese package insert
- Unknown: Participants with no information on baseline renal impairment who received sunitinib malate according to Japanese package insert
Arm/Group | With Renal Impairment | Without Renal Impairment | Unknown
Number analyzed (Participants) | 347 | 1322 | 4
Participants | 336 [19.5 to 23.8] | 1260 | 3

7. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events Who Used Concomitant Cytochrome P450 3A4 (CYP3A4) Inhibitors
Description: A treatment-related adverse event was any untoward medical occurrence attributed to sunitinib malate in a participant who received sunitinib malate. Relatedness to sunitinib malate was assessed by the investigator and sponsor (Pfizer Japan Inc.). A total of 38 drugs including tofisopam, bromocriptin mesilate, and fluvoxamine maleate were defined as CYP3A4 inhibitors.
Time Frame: MAX 2 Years
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- With Concomitant CYP3A4 Inhibitors (Start of Treatment): Participants with concomitant CYP3A4 inhibitors at start of sunitinib malate treatment according to Japanese package insert
- With Concomitant CYP3A4 Inhibitors (During Treatment): Participants with concomitant CYP3A4 inhibitors during sunitinib malate treatment according to Japanese package insert
- Without Concomitant CYP3A4 Inhibitors: Participants without concomitant CYP3A4 inhibitors on sunitinib malate treatment according to Japanese package insert
Arm/Group | With Concomitant CYP3A4 Inhibitors (Start of Treatment) | With Concomitant CYP3A4 Inhibitors (During Treatment) | Without Concomitant CYP3A4 Inhibitors
Number analyzed (Participants) | 82 | 45 | 1546
Participants | 82 [19.5 to 23.8] | 45 | 1472

8. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events Who Were Under Long-Term Treatment
Description: A treatment-related adverse event was any untoward medical occurrence attributed to sunitinib malate in a participant who received sunitinib malate. Relatedness to sunitinib malate was assessed by the investigator and sponsor (Pfizer Japan Inc.). The long-term treatment was defined as the treatment continued more than 24 weeks.
Time Frame: MAX 2 Years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 1673
Participants | 4 [19.5 to 23.8]

9. Secondary Outcome: Numbers of Participants With Treatment-Related Adverse Events Corresponded to Items for Priority Investigation
Description: The following adverse events were defined as items for priority investigation : (1) lung disorder including interstitial pneumonia, (2) bone marrow depression including platelets decreased, white blood cell decreased, and anaemia, (3) haemorrhage including those due to tumor degeneration or shrinkage, (4) cardiac function disturbance including QT interval prolonged and left ventricular ejection fraction decreased, (5) dysfunction adrenal, (6) pancreatic dysfunction including lipase increased, (7) thyroid function decreased, (8) cutaneous symptoms (hand and foot syndrome), (9) serious infections, (10) rhabdomyolysis, myopathy, and (11) reversible posterior leukoencephalopathy syndrome (RPLS). Relatedness to sunitinib malate was assessed by the investigator and sponsor (Pfizer Japan Inc.).
Time Frame: MAX 2 Years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 1673
Participants
  Lung disorder | 19 [19.5 to 23.8]
  Bone marrow depression | 1294
  Haemorrhage | 287
  Cardiac function disturbance | 61
  Dysfunction adrenal | 6
  Pancreatic dysfunction | 313
  Thyroid function decreased | 700
  Cutaneous symptoms (hand and foot syndrome) | 629
  Serious infections | 63
  Rhabdomyolysis, myopathy | 24
  RPLS | 3

10. Other Pre Specified Outcome: Number of Participants With Treatment-Related Serious Adverse Events
Description: A treatment-related adverse event was any untoward medical occurrence attributed to sunitinib malate in a participant who received sunitinib malate. A treatmen-trelated serious adverse event was a treatment-related adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; lifethreatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Relatedness to sunitinib malate was assessed by the investigator and sponsor (Pfizer Japan Inc.).
Time Frame: MAX 2 Years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 1673
Participants | 793

11. Other Pre Specified Outcome: Number of Participants With Treatment-Related Adverse Events Unexpected From Japanese Package Insert
Description: A treatment-related adverse event was any untoward medical occurrence attributed to sunitinib malate in a participant who received sunitinib malate. Relatedness to sunitinib malate was assessed by the investigator and sponsor (Pfizer Japan Inc.). Expectedness of the adverse event was determined according to the Japanese package insert. Relatedness to sunitinib malate was assessed by the investigator and sponsor (Pfizer Japan Inc.).
Time Frame: MAX 2 Years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 1673
Participants | 352 [19.5 to 23.8]

12. Other Pre Specified Outcome: Number of Participants With Treatment-Related Adverse Events Grade 3 or Higher in Common Toxicity Criteria for Adverse Events (CTCAE)
Description: A treatment-related adverse event was any untoward medical occurrence attributed to sunitinib malate in a participant who received sunitinib malate. Relatedness to sunitinib malate was assessed by the investigator and sponsor (Pfizer Japan Inc.). The severity for each adverse event was assessed according to CTCAE as follows: grade 3, severe or medically significant but not immediately life-threatening, hospitalization or prolongation of hospitalization indicated, or disabling; grade 4, life-threatening consequences or urgent intervention indicated; grade 5, death related to adverse event.
Time Frame: MAX 2 Years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 1673
Participants | 1194 [19.5 to 23.8]

ADVERSE EVENTS:
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Sunitinib Malate
Serious Adverse Events (participants affected / at risk) | 1000/1673
Other Adverse Events (participants affected / at risk) | 1530/1673
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib Malate (N=1673)
Anaemia (Blood and lymphatic system disorders) | 56
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 24
Eosinophilia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 8
Lymphopenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 18
Pancytopenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 48
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1
Bone marrow failure (Blood and lymphatic system disorders) | 29
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Atrioventricular block (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 6
Cardiac failure congestive (Cardiac disorders) | 4
Cardio-respiratory arrest (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 3
Sinus bradycardia (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 1
Left ventricular dysfunction (Cardiac disorders) | 2
Cardiac disorder (Cardiac disorders) | 1
Adrenal haemorrhage (Endocrine disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Adrenocortical insufficiency acute (Endocrine disorders) | 2
Hyperthyroidism (Endocrine disorders) | 6
Hypothyroidism (Endocrine disorders) | 52
Thyroid disorder (Endocrine disorders) | 2
Thyroiditis (Endocrine disorders) | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1
Myxoedema (Endocrine disorders) | 1
Vision blurred (Eye disorders) | 1
Vitreous haemorrhage (Eye disorders) | 2
Ulcerative keratitis (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Ascites (Gastrointestinal disorders) | 4
Colitis ulcerative (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 26
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Duodenal perforation (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastric perforation (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 2
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 18
Gastrointestinal perforation (Gastrointestinal disorders) | 5
Gingival bleeding (Gastrointestinal disorders) | 1
Glossitis (Gastrointestinal disorders) | 1
Glossodynia (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 7
Ileus paralytic (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 4
Intestinal perforation (Gastrointestinal disorders) | 5
Large intestine perforation (Gastrointestinal disorders) | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 3
Mouth haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 18
Oesophageal ulcer (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 2
Pancreatic enzyme abnormality (Gastrointestinal disorders) | 7
Pancreatitis (Gastrointestinal disorders) | 2
Pancreatitis acute (Gastrointestinal disorders) | 1
Parotid gland enlargement (Gastrointestinal disorders) | 1
Peptic ulcer (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2
Rectal ulcer (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 12
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 10
Gastroduodenitis (Gastrointestinal disorders) | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 3
Pneumatosis intestinalis (Gastrointestinal disorders) | 3
Diverticular perforation (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 3
Death (General disorders) | 14
Face oedema (General disorders) | 1
Fatigue (General disorders) | 11
Generalised oedema (General disorders) | 2
Impaired healing (General disorders) | 1
Malaise (General disorders) | 37
Multi-organ failure (General disorders) | 3
Oedema (General disorders) | 8
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 3
Pyrexia (General disorders) | 55
Sudden death (General disorders) | 1
Localised oedema (General disorders) | 1
General physical health deterioration (General disorders) | 2
Induration (General disorders) | 1
Disease progression (General disorders) | 187
Bile duct stone (Hepatobiliary disorders) | 1
Cholangitis (Hepatobiliary disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 5
Cholecystitis acute (Hepatobiliary disorders) | 6
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 3
Hepatic function abnormal (Hepatobiliary disorders) | 45
Hyperbilirubinaemia (Hepatobiliary disorders) | 2
Jaundice (Hepatobiliary disorders) | 2
Liver disorder (Hepatobiliary disorders) | 4
Bile duct obstruction (Hepatobiliary disorders) | 1
Drug-induced liver injury (Hepatobiliary disorders) | 2
Acute tonsillitis (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Epididymitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gingivitis (Infections and infestations) | 6
Hepatitis infectious (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 4
Infection (Infections and infestations) | 10
Liver abscess (Infections and infestations) | 1
Lung abscess (Infections and infestations) | 1
Periodontitis (Infections and infestations) | 3
Pharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 27
Postoperative wound infection (Infections and infestations) | 1
Pseudomembranous colitis (Infections and infestations) | 1
Pulmonary tuberculosis (Infections and infestations) | 2
Pyelonephritis (Infections and infestations) | 2
Pyelonephritis acute (Infections and infestations) | 1
Sepsis (Infections and infestations) | 5
Septic shock (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 2
Streptococcal sepsis (Infections and infestations) | 1
Peritonsillitis (Infections and infestations) | 1
Appendiceal abscess (Infections and infestations) | 1
Enteritis infectious (Infections and infestations) | 2
Neutropenic infection (Infections and infestations) | 3
Pneumonia bacterial (Infections and infestations) | 3
Cholecystitis infective (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Alveolar osteitis (Infections and infestations) | 1
Infectious pleural effusion (Infections and infestations) | 2
Peritonitis (Infections and infestations) | 7
Accident (Injury, poisoning and procedural complications) | 1
Brain herniation (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 3
Femur fracture (Injury, poisoning and procedural complications) | 2
Humerus fracture (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 3
Brain contusion (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 15
Aspartate aminotransferase increased (Investigations) | 19
Blood albumin decreased (Investigations) | 1
Blood bilirubin increased (Investigations) | 3
Blood creatine phosphokinase increased (Investigations) | 4
Blood creatinine increased (Investigations) | 15
Blood lactate dehydrogenase increased (Investigations) | 2
Blood potassium increased (Investigations) | 2
Blood pressure decreased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Blood sodium decreased (Investigations) | 1
Blood thyroid stimulating hormone increased (Investigations) | 2
Blood urea increased (Investigations) | 1
Blood uric acid increased (Investigations) | 3
C-reactive protein increased (Investigations) | 7
Electrocardiogram T wave inversion (Investigations) | 1
Haemoglobin decreased (Investigations) | 15
Lipase increased (Investigations) | 19
Lymphocyte count decreased (Investigations) | 10
Neutrophil count decreased (Investigations) | 54
Platelet count decreased (Investigations) | 334
Prothrombin time prolonged (Investigations) | 1
Weight increased (Investigations) | 1
White blood cell count decreased (Investigations) | 95
Ejection fraction decreased (Investigations) | 13
Blood creatine phosphokinase BB increased (Investigations) | 1
Protein urine present (Investigations) | 1
Troponin increased (Investigations) | 1
Cardiac function test abnormal (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 7
Hepatic enzyme increased (Investigations) | 1
Pancreatic enzymes increased (Investigations) | 2
Cell marker increased (Investigations) | 1
Amylase increased (Investigations) | 11
Acidosis (Metabolism and nutrition disorders) | 1
Cachexia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 9
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Fluid retention (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 10
Hyperkalaemia (Metabolism and nutrition disorders) | 12
Hyperuricaemia (Metabolism and nutrition disorders) | 6
Hypoalbuminaemia (Metabolism and nutrition disorders) | 10
Hypocalcaemia (Metabolism and nutrition disorders) | 3
Hyponatraemia (Metabolism and nutrition disorders) | 19
Hypophosphataemia (Metabolism and nutrition disorders) | 3
Hypoproteinaemia (Metabolism and nutrition disorders) | 2
Tumour lysis syndrome (Metabolism and nutrition disorders) | 2
Feeding disorder (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 44
Hyperlipidaemia (Metabolism and nutrition disorders) | 2
Hyperamylasaemia (Metabolism and nutrition disorders) | 1
Hypophagia (Metabolism and nutrition disorders) | 3
Hyperlipasaemia (Metabolism and nutrition disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
Pleural neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 23
Altered state of consciousness (Nervous system disorders) | 8
Cerebellar haemorrhage (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 15
Cerebral infarction (Nervous system disorders) | 9
Depressed level of consciousness (Nervous system disorders) | 3
Diplegia (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 4
Dizziness postural (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 2
Encephalopathy (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Guillain-Barre syndrome (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Hemiparesis (Nervous system disorders) | 1
Hemiplegia (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 1
Intracranial pressure increased (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Monoplegia (Nervous system disorders) | 2
Myasthenia gravis (Nervous system disorders) | 1
Myoclonus (Nervous system disorders) | 1
Nervous system disorder (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Paraplegia (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Brain oedema (Nervous system disorders) | 3
Balance disorder (Nervous system disorders) | 1
VIIth nerve paralysis (Nervous system disorders) | 1
Lacunar infarction (Nervous system disorders) | 1
Metabolic encephalopathy (Nervous system disorders) | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 3
Seizure (Nervous system disorders) | 1
Completed suicide (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Mood swings (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 2
Nephrosclerosis (Renal and urinary disorders) | 1
Nephrotic syndrome (Renal and urinary disorders) | 5
Proteinuria (Renal and urinary disorders) | 4
Renal disorder (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Renal haemorrhage (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 2
Haemorrhage urinary tract (Renal and urinary disorders) | 2
Postrenal failure (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 22
Bladder tamponade (Renal and urinary disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 5
Scrotal ulcer (Reproductive system and breast disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 7
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 16
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 26
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 2
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 24
Purpura (Skin and subcutaneous tissue disorders) | 1
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 5
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2
Aortic dissection (Vascular disorders) | 3
Circulatory collapse (Vascular disorders) | 2
Flushing (Vascular disorders) | 1
Hypertension (Vascular disorders) | 55
Hypotension (Vascular disorders) | 1
Shock (Vascular disorders) | 1
Venous thrombosis (Vascular disorders) | 1
Aneurysm ruptured (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Vascular insufficiency (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 5
Artery dissection (Vascular disorders) | 1
Haematocrit decreased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib Malate (N=1673)
Anaemia (Blood and lymphatic system disorders) | 170
Thrombocytopenia (Blood and lymphatic system disorders) | 109
Hypothyroidism (Endocrine disorders) | 589
Constipation (Gastrointestinal disorders) | 102
Diarrhoea (Gastrointestinal disorders) | 284
Nausea (Gastrointestinal disorders) | 153
Stomatitis (Gastrointestinal disorders) | 285
Malaise (General disorders) | 176
Oedema (General disorders) | 91
Pyrexia (General disorders) | 211
Hepatic function abnormal (Hepatobiliary disorders) | 163
Aspartate aminotransferase increased (Investigations) | 91
Haemoglobin decreased (Investigations) | 85
Lipase increased (Investigations) | 179
Neutrophil count decreased (Investigations) | 176
Platelet count decreased (Investigations) | 694
White blood cell count decreased (Investigations) | 464
Amylase increased (Investigations) | 120
Decreased appetite (Metabolism and nutrition disorders) | 196
Dysgeusia (Nervous system disorders) | 139
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 105
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 603
Rash (Skin and subcutaneous tissue disorders) | 103
Hypertension (Vascular disorders) | 551
Bone marrow failure (Blood and lymphatic system disorders) | 54
Leukopenia (Blood and lymphatic system disorders) | 50
Neutropenia (Blood and lymphatic system disorders) | 23
Hyperthyroidism (Endocrine disorders) | 40
Thyroid disorder (Endocrine disorders) | 23
Eyelid oedema (Eye disorders) | 24
Abdominal discomfort (Gastrointestinal disorders) | 38
Abdominal pain (Gastrointestinal disorders) | 19
Abdominal pain upper (Gastrointestinal disorders) | 22
Cheilitis (Gastrointestinal disorders) | 27
Dyspepsia (Gastrointestinal disorders) | 47
Gastritis (Gastrointestinal disorders) | 52
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 19
Gingival bleeding (Gastrointestinal disorders) | 20
Vomiting (Gastrointestinal disorders) | 79
Pancreatic enzyme abnormality (Gastrointestinal disorders) | 29
Gastric ulcer (Gastrointestinal disorders) | 27
Face oedema (General disorders) | 44
Fatigue (General disorders) | 73
Oedema peripheral (General disorders) | 31
Liver disorder (Hepatobiliary disorders) | 22
Alopecia (Skin and subcutaneous tissue disorders) | 19
Eczema (Skin and subcutaneous tissue disorders) | 18
Erythema (Skin and subcutaneous tissue disorders) | 23
Pruritus (Skin and subcutaneous tissue disorders) | 18
Skin discolouration (Skin and subcutaneous tissue disorders) | 25
Skin disorder (Skin and subcutaneous tissue disorders) | 24
Yellow skin (Skin and subcutaneous tissue disorders) | 57
C-reactive protein increased (Investigations) | 25
Alanine aminotransferase increased (Investigations) | 64
Lymphocyte count decreased (Investigations) | 39
Ejection fraction decreased (Investigations) | 19
Blood pressure increased (Investigations) | 31
Blood alkaline phosphatase increased (Investigations) | 38
Blood creatinine increased (Investigations) | 55
Blood creatine phosphokinase increased (Investigations) | 21
Blood bilirubin increased (Investigations) | 18
Blood thyroid stimulating hormone increased (Investigations) | 51
Blood lactate dehydrogenase increased (Investigations) | 23
Hyperkalaemia (Metabolism and nutrition disorders) | 23
Hyperuricaemia (Metabolism and nutrition disorders) | 65
Hypoalbuminaemia (Metabolism and nutrition disorders) | 19
Hyponatraemia (Metabolism and nutrition disorders) | 20
Headache (Nervous system disorders) | 37
Cough (Respiratory, thoracic and mediastinal disorders) | 26
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 27
Insomnia (Psychiatric disorders) | 51
Gingivitis (Infections and infestations) | 30
Nasopharyngitis (Infections and infestations) | 25
Periodontitis (Infections and infestations) | 23
Pneumonia (Infections and infestations) | 19
Back pain (Musculoskeletal and connective tissue disorders) | 30
Haematuria (Renal and urinary disorders) | 22
Renal impairment (Renal and urinary disorders) | 64
Proteinuria (Renal and urinary disorders) | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.